CLINICAL TRIAL: NCT02984059
Title: A Pilot Study Assessing Risk Factors for Abdominal Pain in Children With Inflammatory Bowel Disease: The ALLAY Study
Brief Title: Study Assessing Risk Factors for Abdominal Pain in Children With Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: Connecticut Children's Medical Center (Other)
Responsible Party: Principal Investigator, Victoria Grossi, Pediatric Fellow/GI Department, Connecticut Children's Medical Center
Other Study IDs: The ALLAY Study
Record Dates: First submitted 2016-02-03; First posted 2016-12-06 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — DNA Probes; Microbiota; Leukocyte L1 Antigen Complex

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — pending
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- IBD w/abdominal pain: Patients with IBD with abdominal pain. Extra colonic biopsies for RNA analysis. If blood and stool samples are collected for standard of care:blood analyzed for both genomic DNA and calprotectin, and stool analyzed for microbiome. If no blood is drawn then a buccal swab done for the genomic DNA analysis and stool analyzed for calprotectin.
  Pain questionnaires:
  Pain Frequency-Severity-Duration Scale Pain Catastrophizing Scale-Child Version Pain Burden Interview Pediatric Quality of Life Inventory Adolescent Pediatric Pain Tool Anxiety/Depression Questionnaires Revised Children's Anxiety and Depression Scale Children's Somatization Inventory Adult Responses to Children's Symptoms
  Interventions: Genetic: Genomic DNA; Genetic: RNA analysis; Genetic: Microbiome; Other: Calprotectin; Other: Pain questionnaires; Other: Anxiety/Depression Questionnaires
- IBD w/out abdominal pain: Patients with IBD and no abdominal pain. Colonoscopy done for standard of care, extra colonic biopsies for RNA analysis. If blood and stool samples are collected for standard of care:blood analyzed for genomic DNA and calprotectin and stool analyzed for microbiome. If no blood is drawn then a buccal swab for the genomic DNA analysis and stool analyzed for calprotectin.
  Pain questionnaires:
  Pain Frequency-Severity-Duration Scale Pain Catastrophizing Scale-Child Version Pain Burden Interview Pediatric Quality of Life Inventory Adolescent Pediatric Pain Tool Anxiety/Depression Questionnaires Revised Children's Anxiety and Depression Scale Children's Somatization Inventory Adult Responses to Children's Symptoms
  Interventions: Genetic: Genomic DNA; Genetic: RNA analysis; Genetic: Microbiome; Other: Calprotectin; Other: Pain questionnaires; Other: Anxiety/Depression Questionnaires
- Colonoscopy other reasons no abd pain: Patients who have a colonoscopy for other reasons, rectal bleeding or polyp surveillance, no abdominal pain. Extra colonic biopsies for RNA analysis. If blood and stool samples are collected for standard of care:blood analyzed for genomic DNA and calprotectin and stool analyzed for microbiome. If no blood is drawn then a buccal swab for the genomic DNA analysis and stool analyzed for calprotectin.
  Interventions: Genetic: Genomic DNA; Genetic: RNA analysis; Genetic: Microbiome; Other: Calprotectin

INTERVENTIONS:
Genetic: Genomic DNA — blood draw
Genetic: RNA analysis — Mucosal Biopsy via colonoscopy
Genetic: Microbiome — Stool microbiome
Other: Calprotectin — stool or blood analysis for calprotectin
Other: Pain questionnaires — PSDS PCS-C/P PBI APPT
  Groups: IBD w/abdominal pain; IBD w/out abdominal pain
Other: Anxiety/Depression Questionnaires — RCADS-25 CSI-24 ARCS
  Groups: IBD w/abdominal pain; IBD w/out abdominal pain

SUMMARY:
To characterize persistent abdominal pain in children with inflammatory bowel disease (IBD) by examining factors such as disease type, activity and location, psychosocial factors, and genetics.

The investigators hypothesize that by using patient pain and psychological assessments in addition to analysis of blood, stool and colonic biopsies, we can better characterize factors that predispose children and adolescents with IBD to have persistent and/or disproportionate abdominal pain.

DETAILED DESCRIPTION:
This is a prospective longitudinal inception cohort pilot study. The study will hopefully provide information about why there is persistent abdominal pain in children with IBD by examining factors such as disease type, activity and location, psychosocial factors, and genetics. Fifty newly diagnosed pediatric IBD patients, age 8-17 years will be enrolled into the study. There will be 2 control groups as well: pain control population: 20 patients with irritable bowel syndrome (IBS) or functional abdominal pain (FAP) diagnosis who have no evidence of bowel inflammation will serve as a pain control population for patients with no active inflammation. To serve as a control population for patients with no abdominal pain or inflammation, the investigators will include 10 patients with no gastrointestinal symptoms, who undergo colonoscopy for various reasons such as painless rectal bleeding, polyp surveillance, etc. The investigators anticipate completing enrollment in 12 months and allowed another 12 months for follow-up.

The study participants will be seen every 3 months for a year and they will have the following procedures/test performed:

1. Standard of care blood and stool samples
2. Pediatric Ulcerative Colitis Activity Index (PUCAI) or Pediatric Crohn's Disease Activity Index (PCDAI)

They will have an endoscopy performed at diagnosis then at 12 months from enrollment.

A magnetic resonance enterography (MRE) will be done at diagnosis.

The following pain and anxiety tests will be performed throughout the study:

Pain:

Pain Severity Duration Scale (PSDS) Pediatric Catastrophizing Scale-Child/Parents (PCS-C/P) Pain Burden Interview (PBI) Adolescent Pediatric Pain Tool (APPT)

Anxiety:

Revised Children's Anxiety and Depression Scale (RCADS-25) Children's Somatization Index (CSI-24) Adult Responses to Children's Symptoms (ARCS)

Blood, rectal biopsies and stool specimens will be obtained throughout various time points of the study to look at hematology, sed rates, C-reactive protein, genomic DNA, colon RNA, stool microbiome and stool calprotectin.

In summary, the investigators will be examining:

1. Relationship between clinical factors and persistent abdominal pain in patients with IBD

   1. Disease type
   2. Location of disease at diagnosis
   3. Extent of disease at diagnosis
   4. Markers of inflammation at diagnosis and over the course of follow up
   5. Active disease vs. inactive disease over the course of follow up
2. Relationship between psychosocial factors persistent abdominal pain, and remission status, specifically in patients with:

   1. Inactive IBD vs. active IBD
   2. Inactive IBD vs. IBS/FAP
   3. We will compare the parental report to patient report in the above mentioned groups
3. Relationship between gene expression, microbiome, persistent abdominal pain, and remission status, specifically in patients with:

   1. Inactive IBD vs. active IBD
   2. Inactive IBD vs. IBS/FAP
   3. Inactive IBD vs. controls with no abdominal pain

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 8 years or < 18 years (achieved 8th birthday but not yet their 18th birthday)
* IBD established by standard criteria
* Anticipated availability for follow up for ≥ 1 year
* Informed consent/assent

Exclusion Criteria:

* Prior abdominal surgery unrelated to IBD
* Active gastrointestinal infection at time of diagnosis (e.g., C. difficile)
* Other co-morbidities that contribute to abdominal pain (e.g., Familial Mediterranean Fever, metabolic disease)
* Preexisting chronic pain disorder (e.g., fibromyalgia)

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study participants will be recruited from the GI clinic here at Connecticut Children's Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2015-10-21 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Changes in abdominal pain from baseline at 3, 6, 9, and 12 months will be assessed using questionnaires | Assessed at baseline then at months 3, 6, 9, and 12
  Changes in abdominal pain from baseline then assessed again at 3, 6, 9, and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Grossi, DO, Principal Investigator — Connecticut Children's Medical Center
Locations (1):
- CT Children's Medical Center, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grossi V, Hyams JS, Glidden NC, Knight BE, Young EE. Characterizing Clinical Features and Creating a Gene Expression Profile Associated With Pain Burden in Children With Inflammatory Bowel Disease. Inflamm Bowel Dis. 2020 Jul 17;26(8):1283-1290. doi: 10.1093/ibd/izz240. PMID 31627210